CLINICAL TRIAL: NCT05499819
Title: The Effect of Beans Compared to Beef on Satiety and Food Intake in Older Adults
Brief Title: Effect of Beans Compared to Beef on Satiety in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Ontario Bean Growers (Unknown)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: REB-22-03-028
Record Dates: First submitted 2022-06-13; First posted 2022-08-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Older Adults
Keywords: beans; beef; satiety; appetite; food intake; energy intake; older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Black beans (Experimental): Canned black beans, drained and rinsed
  Interventions: Other: Canned black beans, drained and rinsed
- Red kidney beans (Experimental): Canned red kidney beans, drained and rinsed
  Interventions: Other: Canned red kidney beans, drained and rinsed
- Extra-lean ground beef (Experimental): Extra-lean ground beef, pan-fried
  Interventions: Other: Extra-lean ground beef

INTERVENTIONS:
Other: Canned black beans, drained and rinsed — Canned black beans, drained and rinsed and consumed in a tortilla wrap
  Arms: Black beans
Other: Canned red kidney beans, drained and rinsed — Canned red kidney beans, drained and rinsed, drained and rinsed and consumed in a tortilla wrap
  Arms: Red kidney beans
Other: Extra-lean ground beef — Extra-lean ground beef, pan-fried and consumed in a tortilla wrap
  Arms: Extra-lean ground beef

SUMMARY:
This human clinical trial is using a randomized crossover design to examine the effect of two varieties of beans compared to beef on satiety and food intake in older adults.

DETAILED DESCRIPTION:
This human clinical trial is using a randomized crossover design that includes 3 study visits separated by washout periods of at least 1 week. Each study visit will last approximately 4 hours and will occur at the Human Nutraceutical Research Unit (HNRU) at the University of Guelph. Study visits will occur in the morning and begin with measurement of fasting body weight. Participants will then complete a baseline satiety questionnaire before they consume a breakfast test meal (that includes either red kidney beans, black beans or extra-lean ground beef). After the breakfast meal, participants will complete a palatability questionnaire. They will also complete more satiety questionnaires at 15, 30, 45, 60, 120, 150 and 180 minutes. After 180 minutes, participants will be consume an ad libitum pizza lunch meal until they are comfortably full. Participants will then be sent home with a food scale and instructions to record everything they eat and drink for the remainder of the day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* ≥60 years old
* BMI between 18.5-30 kg/m2

Exclusion Criteria:

* Medication use that is not at a stable dose (at least 3 months)
* Natural health product use that is not at a stable dose (at least 3 months)
* Antibiotic use in the past 3 months
* Overnight shift work
* Alcohol consumption >14 drinks/week or >4 drinks/sitting
* Anaphylactic food allergy
* Pulse (beans, lentils, chickpeas, dried peas) consumption >4 servings per week
* Recent or intended significant weight loss or weight gain (>4 kg in previous 3 months)
* Breakfast skipping ≥4 days per week
* Vegan diet
* Dislike or unable to consume beans, ground beef, shredded cheddar cheese, white tortilla wraps or frozen cheese pizza
* Three Factor Eating Questionnaire scale scores >11 for Cognitive Restraint, >9 for Disinhibition, and >8 for Hunger
* Diagnosed hypertension (blood pressure >140/90mmHg) that is not managed
* Diagnosed digestive-related condition (i.e. Celiac Disease, constipation, gastritis, gastroesophageal reflux disease, gluten intolerance, hemorrhoids, inflammatory bowel disease (Crohn's, Ulcerative Colitis), irritable bowel syndrome, lactose intolerance)
* Diagnosed cognitive-related condition (i.e. Alzheimer's Disease, amnesia, dementia, generalized anxiety disorder, major depressive disorder, Parkinson's Disease, schizophrenia, traumatic brain injury)
* Medical condition that does not have stable management for at least 3 months
* Medical or surgical event requiring hospitalization in the past 3 months
* Tobacco use
* Cannabis use
* Vape use

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Subjective appetite sensations | Area under the 180 minute curve
  Fullness, satisfaction, hunger, desire to eat, prospective food consumption (measured by a visual analogue scale in mm)

SECONDARY OUTCOMES:
Food intake at an ad libitum pizza meal | 180 minutes after consumption of study treatment (in a breakfast meal)
  Food intake will be measured in grams at an ad libitum cheese pizza lunch meal
24-hour energy intake | 24 hours
  Energy intake measured as kcal for 24 hours after consumption of study treatment (in a breakfast meal) using a weighed food record

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fluit MJ, Adams BF, Ribau ZJ, Duncan AM. Beans Improve Satiety to an Effect that Is Not Significantly Different from Beef in Older Adults: A Randomized, Crossover Trial. J Nutr. 2025 Apr;155(4):1193-1201. doi: 10.1016/j.tjnut.2025.02.008. Epub 2025 Feb 14. PMID 39954740